CLINICAL TRIAL: NCT01307605
Title: Rituximab Plus Lenalidomide or Rituximab Monotherapy for Untreated Patients With Follicular Lymphoma in Need of Therapy. A Randomized, Open-Label, Multicenter Phase II Trial.
Brief Title: Rituximab With or Without Lenalidomide in Treating Patients With Previously Untreated Follicular Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was decided by the trial team to stop the collection of follow up data in trial SAKK 35/10.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 35/10; SWS-SAKK-35-10; 2010-021253-39 (EudraCT Number); CELGENE-SWS-SAKK-35/10 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Active Comparator): Rituximab (MabThera®) will be administered for a maximum of 8 infusions at weeks 1, 2, 3, 4 and again at weeks 12, 13, 14, 15 if the first restaging at week 10 (+/- 1 week) shows a partial response with at least more than 25% reduction in sum of product of diameters
  Interventions: Biological: Rituximab
- Rituximab plus Lenalidomide (Active Comparator): Lenalidomide will be administered as 15 mg flat dose daily, starting 14 days before first and stopping 14 days after last rituximab administration.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Biological: Rituximab — Rituximab (MabThera®) will be administered for a maximum of 8 infusions at weeks 1, 2, 3, 4 and again at weeks 12, 13, 14, 15 if the first restaging at week 10 (+/- 1 week) shows a partial response with at least more than 25% reduction in sum of product of diameters
  Other Names: Rituximab (MabThera)
  Arms: Rituximab
Drug: lenalidomide — Lenalidomide will be administered as 15 mg flat dose daily, starting 14 days before first and stopping 14 days after last rituximab administration.
  Other Names: Lenalidomide (Revlimid)
  Arms: Rituximab plus Lenalidomide

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Lenalidomide may stop the growth of non-Hodgkin lymphoma by blocking blood flow to the cancer. It is not yet known whether rituximab is more effective when given alone or together with lenalidomide in treating patients with follicular lymphoma.

PURPOSE: This randomized phase II trial is studying rituximab to see how well it works compared with giving rituximab together with lenalidomide in treating patients with previously untreated follicular lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the activity of rituximab in combination with lenalidomide versus rituximab alone in patients with previously untreated follicular lymphoma in need of therapy.

Secondary

* To determine the safety of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to grade of disease (grades 1 or 2 vs 3a), presence of bulky disease (defined as masses ≥ 6 cm) (yes vs no), Follicular Lymphoma International Prognostic Index score (1 or 2 vs ≥ 3), and participating centers. Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive rituximab IV on day 1 in weeks 1, 2, 3, 4 and weeks 12, 13, 14, 15 in the absence of disease progression or unacceptable toxicity.
* Arm B: Patients receive rituximab IV as in arm A. Patients also receive oral lenalidomide once daily, starting 14 days before first rituximab administration and last until 14 days after the last rituximab administration, in the absence of disease progression or unacceptable toxicity.

All patients undergo restaging at week 10. Patients who show less than a minimal response (i.e., reduction of more than 25% in sum of product of diameters [SPD]) are off study treatment and transferred to the follow-up phase. Patients undergo a second restaging in week 23.

Some patients may undergo biopsies and blood and bone marrow sample collection periodically for biomarker studies.

After completion of study treatment, patients are followed up periodically for 20 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular lymphoma

  * Stage III or IV disease OR stage II disease not suitable for radiotherapy
  * Grades 1, 2, or 3a disease
* Previously untreated disease
* CD20-positive disease
* Patients in need of systemic therapy, meeting at least 1 of the following criteria:

  * Symptomatic enlarged lymph nodes, spleen, or other lymphoma manifestations
  * Bulky disease ≥ 6 cm in long diameter
  * Clinically significant progression over at least 6 months of any tumor lesion
  * Anemia (hemoglobin < 100 g/L) or thrombocytopenia (platelet count < 100 x 10^9/L) due to lymphoma
  * Clinically significant progressive decrease in hemoglobin or platelet count due to lymphoma
  * B-symptoms, weight loss > 10% within the past 6 months, drenching night sweats, or fever > 38°C not due to infection
* At least one two-dimensionally measurable lesion with longest transverse diameter > 10 mm
* Paraffin-embedded tumor tissue available
* No known CNS involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* EF ≥ 50% for patients with a history of cardiac disease or older than 70 years
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless due to Gilbert syndrome)
* ALT ≤ 2.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 4 weeks prior to, during, and for 12 months after completion of study therapy
* Must be compliant and geographically proximal to allow for proper staging and follow-up
* No serious underlying medical condition, at the judgment of the investigator, which could impair the ability of the patient to participate in the trial (e.g., active autoimmune disease or uncontrolled diabetes)
* No malignancy within the past 3 years except for adequately treated carcinoma in situ of the cervix or localized nonmelanoma skin cancer
* No psychiatric disorder precluding understanding information of trial-related topics, giving informed consent, or interfering with compliance for oral drug intake
* No known hypersensitivity to trial drugs or hypersensitivity to any other components of the trial drugs
* No known HIV positivity or hepatitis C infection
* No serological evidence of current or past hepatitis B infection, unless the serological findings are clearly due to vaccination

PRIOR CONCURRENT THERAPY:

* No prior systemic therapy for this disease
* At least 3 months since prior radiotherapy
* At least 30 days since prior treatment in another clinical trial
* At least 4 weeks since prior and no concurrent corticosteroids unless administered as prophylaxis in at-risk patients for ≤ 3 days or at a dose equivalent to prednisone ≤ 15 mg/day, for indications other than lymphoma or lymphoma-related symptoms
* No concomitant drugs contraindicated for use with the trial drugs
* No other concurrent experimental drugs or anticancer therapy
* No other concurrent investigational treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) | at week 23
  The evaluation of CR is outlined in Appendix 1 Criteria for Evaluation of Response in Non-Hodgkin's Lymphoma.

SECONDARY OUTCOMES:
Best overall response (OR) | within 24 weeks
  OR is defined as either:
  * the disappearance of all evidence of disease (CR or CRu)
  * the regression of measurable disease with no new sites (PR)
Best Overall response (OR) | within 12 weeks
  OR is defined as either:
  * the disappearance of all evidence of disease (CR or CRu)
  * the regression of measurable disease with no new sites (PR)
Progression-free survival | until disease progression, for up to 10 years after randomization
  PFS will be calculated from randomization until the first event of interest:
  * disease progression or relapse according to criteria of Cheson et a.l 1999
  * death from any cause
Time to first off-trial anti-lymphoma therapy | until off-trial therapy administration, for up to 10 years after randomization
  This will be calculated from randomization until the start of the first off-trial anti-lymphoma treatment.
  Patients not receiving any off-trial anti-lymphoma treatment will be censored at the last follow-up visit.
Overall survival | every 6 months for up to 10 years after randomization
  OS will be calculated from randomization until death. Patients not experiencing an event will be censored at the last date they were known to be alive.
Adverse events, including laboratory abnormality assessments and vital signs | from inclusion until 30 days after treatment discontinuation
  This will be evaluated using the NCI CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Zucca, MD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni; Eva K. Kimby, MD, PhD, Study Chair — Karolinska Institutet; Felicitas Hitz, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Bjorn Ostenstad, MD, Principal Investigator — Ullevaal University Hospital
Locations (33):
- Norway (6):
  - Haukeland Hospital - University of Bergen, Bergen
  - Sorlandet Sykehus HF Kristiansand, Kristiansand
  - Ullevaal University Hospital, Oslo
  - Helse Stavanger HF, Stavanger
  - University Hospital of North Norway - Tromso, Tromsø
  - St. Olavs University Hospital, Trondheim
- Sweden (9):
  - Sahlgrenska University Hospital, Gothenburg
  - University Hospital of Linkoping, Linköping
  - Sunderbyn Hospital, Luleå
  - Lund University Hospital, Lund
  - Karolinska University Hospital - Huddinge, Stockholm
  - Karolinska University Hospital - Solna, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Norrlands University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (18):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Oberwallis - Brig, Brig
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - University Hospital, Geneva
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Kantonsspital Winterthur, Winterthur
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menter T, Tzankov A, Zucca E, Kimby E, Hultdin M, Sundstrom C, Beiske K, Cogliatti S, Banz Y, Cathomas G, Karjalainen-Lindsberg ML, Grobholz R, Mazzucchelli L, Sander B, Hawle H, Hayoz S, Dirnhofer S. Prognostic implications of the microenvironment for follicular lymphoma under immunomodulation therapy. Br J Haematol. 2020 May;189(4):707-717. doi: 10.1111/bjh.16414. Epub 2020 Feb 3. PMID 32012230
- [Derived] Zucca E, Rondeau S, Vanazzi A, Ostenstad B, Mey UJM, Rauch D, Wahlin BE, Hitz F, Hernberg M, Johansson AS, de Nully Brown P, Hagberg H, Ferreri AJM, Lohri A, Novak U, Zander T, Bersvendsen H, Bargetzi M, Mingrone W, Krasniqi F, Dirnhofer S, Hayoz S, Hawle H, Vilei SB, Ghielmini M, Kimby E; Swiss Group for Clinical Cancer Research and the Nordic Lymphoma Group. Short regimen of rituximab plus lenalidomide in follicular lymphoma patients in need of first-line therapy. Blood. 2019 Jul 25;134(4):353-362. doi: 10.1182/blood-2018-10-879643. Epub 2019 May 17. PMID 31101627